CLINICAL TRIAL: NCT04377542
Title: Randomized Controlled Trial on Ligation of Intersphincteric Fistula Tract (LIFT) Versus Modified Parks Technique Versus Two-Stage Seton In Treatment of Complex Anal Fistula
Brief Title: RCT on LIFT Versus Modified Parks Technique Versus Two-Stage Seton
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mansoura152020
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Parks, Recreational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LIFT (Active Comparator): Ligation of intersphincteric fistula tract
  Interventions: Procedure: LIFT
- Parks (Active Comparator): Modified Parks technique
  Interventions: Procedure: Parks
- Seton (Active Comparator): Two-stage seton placement
  Interventions: Procedure: Seton

INTERVENTIONS:
Procedure: LIFT — Ligation of the fistula tract in the intersphincteric plane
  Arms: LIFT
Procedure: Parks — Modified Parks fistulotomy with complete internal anal sphincterotomy
  Arms: Parks
Procedure: Seton — Excision of the superficial part of fistula tract and tying loose seton around the remaining part and anal sphincter muscles
  Arms: Seton

SUMMARY:
LIFT is a sphincter-saving procedure that is based on the concept of secure closure of the internal opening and concomitant removal of infected cryptoglandular tissue in the intersphincteric plane. Modified Parks technique involves adequate drainage of the intersphincteric space by extending the internal anal sphincterotomy. Placement of seton in the fistula track has been used for a long time and is still being currently used. Drainage two-stage seton is used to promote adequate drainage of infection and can be employed as a definitive treatment of anal fistula.

This present randomized study aimed to compare LIFT, modified Parks technique, and two-stage seton in treatment of complex anal fistula in terms of success of treatment and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients of either sex aged less than 65 years presenting with complex anal fistula were included. Complex anal fistulas were defined as high trans-sphincteric (involving more than 30% of the external anal sphincter), extra-sphincteric, supra-sphincteric, horse-shoe fistulas and anterior fistulas in females

Exclusion Criteria:

* Patients with simple anal fistula (intersphincteric and low trans-sphincteric anal fistula)
* Patients with associated anorectal pathology such as anal fissure, hemorrhoids, rectal prolapse, neoplasm, solitary rectal ulcer, inflammatory bowel diseases.
* Patients on long-acting steroids or immunosuppressive drugs.
* Patients with fecal incontinence (FI)
* Patients with previous anorectal operations including surgery for previous anal fistula.
* Patients with ASA score (American society of anesthesiologists) of III and higher

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Healing of anal fistula | 6 months after surgery
  complete epithelization of the surgical wound was ascertained, the external and the internal openings were closed, and no discharge was experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No